CLINICAL TRIAL: NCT06944392
Title: Evaluating Pumpkin Seed Oil Extract Supplementation on Bladder Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Julia Geynisman-Tan, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00221825
Record Dates: First submitted 2025-02-04; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-02

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taking pumpkin seed extract (Experimental): Upon a patient's enrollment into the study and completion of initial study questionnaires, a research team member will provide the patient with a single bottle of pumpkin seed oil extract. Enrolled patients will be instructed to initiate using the pumpkin seed oil extract starting the day they receive the supplement. Patients will start taking one pill by mouth per day for 12 weeks. They will also be advised to contact their urogynecologist for follow-up if they have not noticed improvement in their bladder health following 3 months of use. Furthermore, they will be counseled about not starting new medications or supplements during their time as a study participant and not sharing their pumpkin seed oil extract with anyone else during their time as a study participant.
  Interventions: Dietary Supplement: Pumpkin Seed Extract

INTERVENTIONS:
Dietary Supplement: Pumpkin Seed Extract — This is the only intervention

SUMMARY:
This is a pilot study to assess using validated outcome measures how ingesting pumpkin seed oil extract supports patient bladder function in a United States population.

DETAILED DESCRIPTION:
OBJECTIVES:

Null hypothesis - Ingesting 1000mg daily of Cucurbita pepo pumpkin seed oil extract leads to no change in patient-reported bladder function reflected through Lower Urinary Tract Dysfunction Network Symptom Index-10 (LURN-SI) survey scores between their baseline assessment and at 12 weeks of supplement use.

Primary Objective:

1. Assess changes in patient-reported bladder function reflected through their responses on the LURN-SI survey.

Secondary Objectives:

1. Assess rapid changes in patient-reported bladder function reflected through their responses on the LURN-SI survey following 4 weeks of supplement use.
2. Assess changes in patient-reported pelvic floor control reflected through their responses on the Pelvic Pain and Urgency/Frequency (PUF) questionnaire.
3. Assess patient willingness to continue with supplement use via responses on the Medication Adherence Questionnaire (MAQ).
4. Assess for any relationships in changes in patient bladder function or pumpkin seed extract adherence with their experience using complementary and alternative medicine.

BACKGROUND:

Overactive bladder (OAB) describes a change in bladder function with more frequent and urgent trips to the bathroom to urinate that interfere with the patient's quality of life. Patients with OAB experience urinary frequency, urgency, and leakage, and the 2011 EpiLUTS study estimated 33% women in the United States experience bothersome OAB.1 OAB adversely impacts quality-of-life and incurs almost $7 billion USD in healthcare-related costs annually within the United States, with costs being up to 5 times greater for women than men.2-4 The additional costs of items such as continence sanitary products may be prohibitive, which likely disproportionately impacts socially vulnerable patients.5,6 Despite significant efforts previous invested into evaluating causes for OAB and in developing treatments, the exact mechanism for OAB remains poorly understood and the side effects from pharmacologic treatment can be frustrating.

As a result, certain patients opt to manage their OAB through complementary and alternative medicine (CAM).7 This includes use of nutritional supplement products. One study found that one online vendor carried 147 products marketed as supporting bladder health which contained 65 distinct supplements, and over 50% of products listed pumpkin seed extract as an ingredient.8 However, the exact mechanism for how pumpkin seed oil extract supports bladder function remains poorly understood.

Limited animal study data suggest ingestion of pumpkin (Cucurbita) seed oil extract is associated with increased bladder compliance on urodynamic studies and decreased urinary frequency.9,10 It is posited that the high arginine levels found in pumpkin seeds drive nitric oxide production via the arginine nitric oxide pathway which subsequently contribute to findings of bladder relaxation.

The utility of pumpkin seed oil is further explored in the management of benign prostate hypertrophy (BPH)-associated symptomatology. One review noted use of Cucurbita pepo was associated with improvements in BPH symptoms, decreased detrusor activity, and improvements in urodynamic measurements.11 Subsequent studies utilizing Cucurbita pepo similarly described improvements in patient-reported BPH symptoms and nocturia episodes, in residual urine volumes, and in quality-of-life.12,13 A study comparing performance of Cucurbita pepo with Tamsulosin echoed these outcomes.14 Patients using Cucurbita pepo also reported no side effects with use.15 While pumpkin seeds are known to contain properties associated with reductions in dihydrotestosterone levels, it remains unclear how they contribute to these results or whether any of these effects would be observed in women.16

Studies on outcomes with pumpkin seed oil in female patients are limited however. Patients utilizing 10 grams of Cucurbita maxima oil daily for 12 weeks in one study noted improvements in their overactive bladder scores (OAB-SS).17 Meanwhile, a comparison of using a combination of Cucurbita pepo seed extract and soy germ extract versus maltodextrin alone for 12 weeks noted improvements in OAB symptoms with both approaches.18 Another study comparing impact of daily Solifenacin use with daily use of a CAM formulation containing Cucurbita maxima over a 12 week period described improvements in OAB symptoms across both treatment methods, with CAM generating superior results compared to Solifenacin.19 A retrospective study similarly examining daily use of an oral combination supplement containing Cucurbita maxima over 12 weeks described improvements in both bladder function and patient quality-of-life.20

At this time, a number of patients seeking care with Northwestern's Integrated Pelvic Health Program (IPHP) have verbalized desire to utilize more conservative approaches to supporting their bladder function, including initiation of nutritional supplements such as pumpkin seed oil extract. Unfortunately, the previously mentioned studies in female patients were conducted outside of the United States using small sample sizes drawn from populations not representative of the United States' patient population. These studies also varied in use of pumpkin seed oil extract dosages and species, of supplement combinations, and of validated outcome measures. Hence, it is important to re-study how ingestion of pumpkin seed oil extract supports patient bladder function in a United States population using validated outcome measures.

Purpose: To perform a pilot study assessing how ingesting pumpkin seed oil extract supports patient bladder function.

STUDY ENDPOINTS:

At the conclusion of this study, research team members will review participant questionnaire responses to identify any changes in participant bladder function, specifically changes in frequent voiding and sensation of bladder fullness and pressure, following initiation of pumpkin seed oil extract supplement.

Research team members will also assess for any changes in participant pelvic floor control and for participant willingness to continue use of a nutritional supplement marketed to support bladder function.

In addition, participant demographic information will also be reviewed to verify participant population heterogeneity at time of final data analysis for purposes of data generalizability and to draw potential relationships between particular demographic characteristics and participant-reported outcomes.

STUDY INTERVENTION(S) / INVESTIGATIONAL AGENT(S):

Pumpkin (Cucurbita pepo) seed oil extract (NOW brand, 1000mg pumpkin seed oil extract per pill, 100 pills per bottle) will be purchased from an online vendor. Once received, the pumpkin seed oil extract will be stored in a secured cabinet space per manufacturer guidelines. This cabinet will only be accessible to this study's team members.

Upon a patient's enrollment into the study and completion of initial study questionnaires, a research team member will provide the patient with a single bottle of pumpkin seed oil extract. Enrolled patients will be instructed to initiate using the pumpkin seed oil extract starting the day they receive the supplement. Patients will start taking one pill by mouth per day for 12 weeks. They will also be advised to contact their urogynecologist for follow-up if they have not noticed improvement in their bladder health following 3 months of use. Furthermore, they will be counseled about not starting new medications or supplements during their time as a study participant and not sharing their pumpkin seed oil extract with anyone else during their time as a study participant.

PROCEDURES INVOLVED:

Study design:

This is a prospective pilot study assessing how use of pumpkin seed oil extract supplement impacts patient perceptions of bladder function, specifically via changes in frequent voiding and sensation of bladder fullness and pressure. Patients will be recruited from across IPHP offices to ensure sample size can be reached in a reasonable time frame and to help with generalizability of the findings. Patients who report symptoms of overactive bladder at their initial visit with IPHP and desire conservative management strategies may be eligible for this study pending review of study inclusion and exclusion criteria.

Patients desiring conservative management will be counseled on standard care options and will then also be offered information about this study. Patients expressing interest will be informed they will contacted by a research team member for further information about the study. Research team members will review patient charts to ensure compliance with this study's inclusion and exclusion criteria. Patients will then meet with a research team member at their same IPHP visit who will counsel them about the study and discuss their eligibility and potentially enrolling in the study.

Following completion of study enrollment consent forms, participants will complete via REDCap at their same office visit on either their personal electronic device or a device provided research staff the LURN-SI, PUF, MAQ, and patient demographic questionnaires. After completing the questionnaires, they will be issued a bottle of pumpkin seed oil extract and asked to start taking one pill by mouth per day for 12 weeks. They will also be advised to contact their urogynecologist for follow-up if they have not noticed improvement in their bladder health following 3 months of use. Furthermore, they will be counseled about not starting new medications or supplements during their time as a study participant and not sharing their pumpkin seed oil extract with anyone else.

Neither the IPHP healthcare team members (attending physicians, fellow physicians, advanced practice registered nurses) nor patients can be blinded to the intervention. Following initiation of pumpkin seed oil extract supplement, patients will continue receiving standard care from their healthcare team members. They will also be sent via REDCap follow-up questionnaires to complete at 4 weeks and 12 weeks following study enrollment.

This study will also be posted on clinicaltrials.gov.

Sample size

Given lack of data on pumpkin seed oil extract supplementation on bladder function within a United States population, we elected to recruit a feasible sample size of 30 patients to conduct a pilot study.

If we anticipate the rate of participant drop-out or withdrawal from the study to be 33%, we project needing to enroll 40 patients to achieve our desired final sample size.

DATA AND SPECIMEN BANKING

All data will be stored on the secure REDCap (Research Electronic Data Capture) server. The data will be stored there for the duration of the study, including during the period of data analysis and manuscript preparation. Patient-identifying information will be destroyed 2 years following study completion. Only this study's research team members will have access to the study's REDCap file. No specimens will be banked for future use.

Each patient will be assigned a unique identifier number and they will be sent the number via REDCap-generated emails sent to their preferred email address. They will use this unique identifier number for entering responses into REDCAP at time of study enrollment, and at 4 weeks and 12 weeks after initiating pumpkin seed oil extract.

Patient-identifying information will remain stored on REDCap for two years to enable sufficient time for completion of participant response acquisition and for subsequent data analysis. All data will be destroyed at the conclusion of this project.

ELIGIBILITY:
Inclusion Criteria:

* All patients evaluated at Northwestern's IPHP who report bladder function consistent with overactive bladder (urinary urgency, with or without urinary frequency more than 8 times daily or nocturia, with or without urgency urinary incontinence) at their index visit, who are also willing to use a dietary supplement and not initiate additional behavioral, medication or procedural treatment for 12 weeks following pumpkin seed oil extract initiation.

Exclusion Criteria:

* Patients with any of the following will be excluded from the study:
* Use of other supplements that contain pumpkin seed oil
* ≥Stage 3 pelvic organ prolapse
* Urinary post-void residual ≥150cc
* Culture-proven urinary tract infection at time of study enrollment
* Recurrent urinary tract infection
* Neurogenic bladder
* Abdominal or pelvic malignancy
* Initiation of new overactive bladder medications or supplements during study period or in the 3 months immediately preceding study enrollment
* History of surgery in the past 12 months for pelvic organ prolapse, stress urinary incontinence, urgency urinary incontinence, or fecal or flatal incontinence
* Patient's primary language is not English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
LURN-SI | 12 weeks
  Assess changes in patient-reported bladder function reflected through their responses on the LURN-SI survey.

SECONDARY OUTCOMES:
Rapid change in LURN-SI | 4 weeks
  Assess rapid changes in patient-reported bladder function reflected through their responses on the LURN-SI survey following 4 weeks of supplement use.
PUF Questionnaire | 12 weeks
  Assess changes in patient-reported pelvic floor control reflected through their responses on the Pelvic Pain and Urgency/Frequency (PUF) questionnaire.
Supplement Adherence | 12 weeks
  Assess patient willingness to continue with supplement use via responses on the Medication Adherence Questionnaire (MAQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Single institution pilot study. Data will be published in aggregate analysis but individual data will not be shared.